CLINICAL TRIAL: NCT04283214
Title: A Comparison of Cardiopulmonary Resuscitation Outcomes Between Traditional and Endomorphic Manikins
Brief Title: A Comparison of CPR Outcomes Between Traditional and Endomorphic Manikins With and Without Equipment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HE20101
Record Dates: First submitted 2020-01-02; First posted 2020-02-25 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional manikin (Active Comparator): CPR performed on a traditional manikin
  Interventions: Other: Cardiopulmonary Resuscitation
- Traditional manikin with athletic equipment (Experimental): CPR performed on a traditional manikin wearing athletic equipment
  Interventions: Other: Cardiopulmonary Resuscitation
- Bariatric manikin (Experimental): CPR performed on a bariatric manikin
  Interventions: Other: Cardiopulmonary Resuscitation
- Bariatric manikin with athletic equipment (Experimental): CPR performed on a bariatric manikin wearing athletic equipment
  Interventions: Other: Cardiopulmonary Resuscitation

INTERVENTIONS:
Other: Cardiopulmonary Resuscitation — Cardiopulmonary Resuscitation based on 2015 American Heart Association guidelines with and without protective equipment on traditional and endomorphic manikins

SUMMARY:
The study's research design is a randomized experiment. 50 emergency responders (emergency medical responders, emergency medical technicians, advanced emergency medical technicians, and paramedics) will be recruited for this research. All data collection will take place in Lab 14 of the Benson Bunker Fieldhouse or a professional, confidential location of the participant's choosing.

Prior to CPR performance, participants will be given an informed consent form to sign. The form will be explained in detail by the researcher collecting data. After obtaining informed consent, participants will be asked to fill out a demographic questionnaire to collect information such as age, gender, years of emergency responder experience/employment, and years of CPR certification. Demographic information provided by participants will be utilized in data analysis. The demographics form should take approximately five minutes to complete. Participants will be randomly assigned to the four trials they will partake in and instructed via oral script (one for over and one for under football shoulder pads) to perform four-trials total of three-minute single-rescuer CPR on both a traditional CPR manikin and "Fat Old Fred" (bariatric) CPR manikin. CPR must be performed in accordance with the American Heart Association's 2015 CPR Guidelines and participants will use a CPRmeter 2 device to collect data to determine the quality of CPR components (chest compression depth/recoil, compression rate, CPR compression duration, mean depth, mean rate, and total number of compressions). The entire study session should take 25 to 30 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Emergency responders employed through the ambulance stations located in North Dakota and Minnesota
* Current CPR/first-aid certification
* Active clinician, educator, or administrator.

Exclusion Criteria:

* Cardiovascular conditions inhibiting CPR performance
* Respiratory conditions inhibiting CPR performance
* Musculoskeletal conditions inhibiting CPR performance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Compression depth % | 2 minutes
  percent of time chest is compressed to adequate depth
Compression rate | 2 minutes
  number of compressions per minute
Chest recoil | 2 minutes
  percent of time chest fully recoils
Compression depth | 2 minutes
  average depth of compressions
Compression rate % | 2 minutes
  percent of time compressions are performed at an adequate rate

CONTACTS AND LOCATIONS:
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No